CLINICAL TRIAL: NCT05531019
Title: COVID-19 Sequelae: Treatment and Monitoring of Persistent Symptoms, a Decentralized Approach Focus on the Patient. Use of Dietary Supplement Based on Sea Urchin Eggs With Echinochroma A.
Brief Title: COVID-19 Sequelae: Treatment and Monitoring. A Dietary Supplement Based on Sea Urchin Eggs With Echinochroma A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fernando Saldarini (Other)
Collaborators: Universidad Nacional de la Patagonia San Juan Bosco (Unknown); Ministerio de Ciencia, Tecnologia e Innovación, Argentina (Unknown); Hospital de Infecciosas Francisco Javier Muniz (Other Government)
Responsible Party: Sponsor-Investigator, Fernando Saldarini, Head of Neumology, Hospital Donación Francisco Santojanni
Organization: Hospital Donación Francisco Santojanni (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5832
Record Dates: First submitted 2022-08-19; First posted 2022-09-07 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Long COVID
Keywords: Covid-19; sequalae; long covid; lung; telemedicine; brain; biomarker
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — echinochrome A

STUDY DESIGN:
Intervention Model Description: Ramdomized Control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The vials of the nutraceutical are identical to each other as well as the labels. It is impossible to distinguish one from the other.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Supplement with sea urchin egg extract (Experimental): Ingestion of dietary supplement with 0,025% of Echinochrome A (ingested 3ml twice a day for 90 days), 1,5mg daily consumption from sea urchin egg extract (Arbacia dufresnii)
  Interventions: Dietary Supplement: Echinochrome A
- Control (Placebo Comparator): Ingestion of 3ml twice a day for 90 days of placebo
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Echinochrome A — Dietary Supplement with Echinochroma A Simple randomized design, in this arm patients will take 6ml of a 0.025% Echinochroma A solution twice a day for 90 days. 3 mg of Echinochroma A will be consumed per day.
  Other Names: EchA Marine
  Arms: Dietary Supplement with sea urchin egg extract
Other: Control — Simple randomized design, in this arm patients will take 6ml of an fructose aqueous solution twice a day for 90 days with the same flavor as the treatment
  Arms: Control

SUMMARY:
The aim of this study is to assess the efficacy and efficiency of a nutraceutical from sea urchin eggs with Echinochrome A in the inflammation of tissues in subjects with long Corona Virus (COVID) syndome

DETAILED DESCRIPTION:
This is a double-blind placebo-controlled study in approximately 60 subjects with long COVID syndrome. After being informed about the study and potential risks, all subjects giving written informed consent will be screened to assess initial respiratory, cardiological inflammatory, neurological and emotional conditions. Prior to the first administration of the treatment, subjetcs will be randomized to receive three vials of the Dietary Supplement with sea urchin eggs extract with presence of the antioxidant Echinochrome A or placebo. According with the ACRO suggestions this study is focus on the patients. Subjects will be monitor by a Telemedicine platform called SkyMed developed for this study to assess their health daily and will have a weekly virtual meeting with a counselors to assess emotional state. Subjects will attend tp the Hospital, at the beggining of the study, and after finishing the vials of the Dietary Supplement (30, 60 and 90 days). Clinical, cardiological, neumonological and neurological studies will carried out to asses the systemic health as well as the quality of life indicators. Inflammation, trombolotic and inmune indicators will be assess in blood samples (basal, 30, 60 and 90 days).

The main objetivec behind this clinical trial is to diminish ROS in the cells, enhance gluthation pathways and diminish cellular inflammation. Echinochrome A is a powerfull marine poliphenol with known antioxidant activity found in the eggs, shells and spines of sea urchins, that had been use in eastern medicien for a long time. Powder of sea urchin eggs are mention in Materia Medica back far 1647 as a powerfull anti inflamation agent.

ELIGIBILITY:
Inclusion Criteria:

1. Positive diagnosis of COVID-19 in at least the last 12 weeks
2. Diagnosis of COVID Persistent, COVID sequalea, Long COVID
3. Adult men or non-pregnant adult women between the ages of 18 and 60.
4. The patient (or legally authorized representative) provides your informed consent before initiating any study procedure.
5. The patient (or legally authorized representative) understands and agrees comply with the planned study procedures. 6. Agreement not to participate in another trial ofintervention for the treatment of COVID-19 until day 60 after the start of the trial.

Exclusion Criteria:

* 1. Patients without persistent COVID symptoms. 2. Patients unable to give informed consent. 3. Patients without a positive result for COVID-19. 4. Pregnancy or lactation. 5. In the doctor's opinion, the patient with advanced organ dysfunction that would not make participation appropriate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
Change of symptoms over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) during rutine medical checkup. | Baseline, 4 weeks, 8 weeks, 12 weeks
  Measuring the symptoms as presence o absence of chest pain, cough, headache, sleep disorders, dysgeusia, myalgia, arthralgia.
Change of lung capacity over four times (baseline, 4 weeks, 8 weeks, 12 weeks) assessed during spirometry. | Baseline, 4 weeks, 8 weeks, 12 weeks
  The main variables of forced spirometry that are measured are the forced vital capacity (FVC) and the forced expiratory volume in the first second (FEV1). The FVC represents the maximum volume of air exhaled in a maximal effort expiratory maneuver, initiated after a maximal inspiration maneuver, expressed in liters. FEV1 corresponds to the maximum volume of air exhaled in the first second of the FVC maneuver, also expressed in liters. In turn, the FEV1/FVC ratio shows the relationship between both parameters.
Change of walking distance during a six minutes walk test (6MWT) over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) | Baseline, 4 weeks, 8 weeks, 12 weeks
  The 6MWT is used, among other things, to assess and control cardiovascular and pulmonary performance below the anaerobic threshold. This test is used for the clinical evaluation of the basic motor property endurance and measures the distance a patient can walk as quickly as possible on a flat, hard surface in a period of 6 minutes. It will be measured in meters.
Change of depression measured over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via the Beck Health Questionnaire. | Baseline, 4 weeks, 8 weeks, 12 weeks
  The Beck Anxiety Inventory is a useful tool to assess somatic symptoms of anxiety, both in anxiety disorders and depressive symptoms. The questionnaire consists of 21 questions, providing a score range between 0 and 63.
Change in the quality of life meassured over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via visual analog scale of EuroQol (EQ-VAS). | Baseline, 4 weeks, 8 weeks, 12 weeks
  EQ-VAS which is a scale of 0 to 100 that allows individuals to place themselves according to how they perceive their overall health status (0 is the worst and 100 the best health status)
Presence or absence of Myocarditis meassured over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via electrocardiogram. | Baseline, 4 weeks, 8 weeks, 12 weeks
  Electrocardiographic signs in patients with myocarditis include T-wave and ST-segment abnormalities, ST-segment elevation
Change in the cognitive function meassured over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via Trial Making test (TMT). | Baseline, 4 weeks, 8 weeks, 12 weeks
  The TMT is timed (seconds) and performed in two parts using only a pen and a piece of paper.It can provide insights into a person's cognitive function based on how fast they can search, scan, and process visual information without losing track of what they are doing.The test also provides information about a person's mental flexibility.
Change in the cognitive function meassured over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via Phonological verbal fluency test. | Baseline, 4 weeks, 8 weeks, 12 weeks
  Verbal fluency tests are commonly used to investigate lexical skills and semantic knowledge. for number of words beginning with the letters F, A, and S and for to al number of words beginning with either letter generated per minute.
Change in the cognitive function meassured over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via Frontal assessment battery (FAB). | Baseline, 4 weeks, 8 weeks, 12 weeks
  The Frontal Assessment Battery (FAB) is a cognitive test that incorporates several clinical assessments to screen for frontotemporal dementia (FTD), including S-word generation, similarities, Luria's test, grasp reflex, and the Go-No-Go test.
Change in the cognitive function meassured over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via clock test (CDT). | Baseline, 4 weeks, 8 weeks, 12 weeks
  The CDT is used to quickly assess visuospatial and praxis abilities, and may determine the presence or absence of both attention and executive dysfunctions: ask the patient to draw the face of a clock and then to draw the hands to indicate a particular time.
Change in the cognitive function meassured over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via Analogies (WAIS-III). | Baseline, 4 weeks, 8 weeks, 12 weeks
  Wais-III is an instrument for assessing Verbal Comprehension, it refers to conceptualization, knowledge and verbal expression. The subject must answer questions that measure practical knowledge, word meanings, reasoning, and the ability to express ideas in words. The Analogies subtest assesses fluid intelligence where the subject's ability to solve new problems that do not depend on schooling or formal culture is reflected: before a series of words presented, the examinee must explain the similarity of common objects or concepts that those terms represent. Maximum direct score 33 points.
Change in the memory over time-points ) baseline, 4 weeks, 8 weeks, 12 weeks) via Rey Auditory Verbal Learning Test. | Baseline, 4 weeks, 8 weeks, 12 weeks
  The test is designed as a list-learning paradigm in which the patient hears a list of 15 nouns and is asked to recall as many words from the list as possible. After five repetitions of free-recall, a second "interference" list (List B) is presented in the same manner, and the participant is asked to recall as many words from List B as possible. After the interference trial, the participant is immediately asked to recall the words from List A, which she or he heard five times previously. After a 20 min delay, the participant is asked to again recall the words from List A. After this "delayed recall" task, a list of 50 words is presented containing all of the words from Lists A. The score given for each trial is the total number of words recalled. Normal scores are 6 words hit on the first trial and 12 or 13 on the fifth trial.
Change in the memory over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via the memory failures of every-day (MFE) | Baseline, 4 weeks, 8 weeks, 12 weeks
  The Memory Failures of Everyday-MFE Questionnaire was used for the subjective assessment of memory. It consists of 28 items on situations and activities of daily living. Each item was scored on a 0-2 point scale ("never or rarely", "sometimes", "many times").
Change in the overall cognitive ability over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) assessed during Addenbrooke's Cognitive Examination Revised (ACE-R) test. | Baseline, 4 weeks, 8 weeks, 12 weeks
  The ACE-R takes between 12 and 20 min (average 16) to administer and score in a clinical setting. It contains 5 sub-scores, each one representing one cognitive domain: attention/orientation (18 points), memory (26 points), fluency (14 points), language (26 points) and visuospatial (16 points). ACE-R maximum score is 100, composed by the addition of the all domains
Change in the overall memory over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) assessed during Digit Span (WAIS-III): Forward. | Baseline, 4 weeks, 8 weeks, 12 weeks
  The Digit Span score is the length of the longest correctly repeated sequence. The idea was to test how much a person can receive, process and remember for a variety of elements. On average a person is not capable of retaining more than 7 pieces of information. This means that when the longest repeated sequence is 7, the participant reached level 7. The test was assessed in forward orders of the digits.
Change in the assess aspects such as selective attention and inhibitory control over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via Stroop test. | Baseline, 4 weeks, 8 weeks, 12 weeks
  Throughout the Stroop test, a total of three different tasks are carried out, through three sheets in which five columns of 20 elements appear. Each one of the tasks is carried out during a certain time (for example, forty-five seconds), scoring the successes for later evaluation. The successes that the subject has had during the test or the time it takes to react to the stimulation are valued, paying attention to what is reflected in each of the sheets or tasks.
Changes in the expression of language over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via Boston Nomination Test. | Baseline, 4 weeks, 8 weeks, 12 weeks
  The Boston vocabulary test consists of 60 figures, ordered from the easiest to the most difficult. The figures are presented in order, allowing the subject 20 seconds to respond. The scores provided by the test are: - The number of correct answers given spontaneously.
Changes in the expression of language over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via semantic Verbal Fluency test. | Baseline, 4 weeks, 8 weeks, 12 weeks
  The Semantic Verbal Fluency (SVF) test entails the generation of words from a given category within a pre-set time of 60 seconds.
Changes in sleep behaviors over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via The Pittsburgh Sleep Quality Index (PSQI) | Baseline, 4 weeks, 8 weeks, 12 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is the most widely used sleep questionnaire in adults, consisting of 24 questions. The first 19 questions are answered by the evaluated person taking into account what they have experienced during the last month.
  Resultados de traducción Sleep quality index (PSQI)
Changes in concussion over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via king figure method. | Baseline, 4 weeks, 8 weeks, 12 weeks
  Demonstration and test cards for the King-Devick test, a candidate rapid sideline screening for concussion based on speed of rapid number naming. To perform the King-Devick test, participants are asked to read the numbers on each card from left to right as quickly as possible, but without making any errors. Following completion of the demonstration card (upper left), subjects are then asked to read each of the three test cards in the same manner. The times required to complete each card are recorded in seconds using a stopwatch. The sum of the three test card time scores constitutes the summary score for the entire test, the King-Devick time score. Numbers of errors made in reading the test cards are also recorded; misspeaks on numbers are recorded as errors only if the subject does not immediately correct the mistake before going on to the next number.
Changes in olfactory-specific quality of life over time-points (baseline, 4 weeñs, 8 weeks, 12 weeks) via questionnaire of olfactory disorders-negative statements (QOD-NS) and a short version of QOD-NS (sQOD-NS). | Baseline, 4 weeks, 8 weeks, 12 weeks
  The QOD-NS questionnaire consists of 17 negative statements about the degree to which patients suffered from olfactory impairment. Patients can agree, partly agree, partly disagree, or disagree in each statement which ranges from 0 to 3. A total score of 0-51 is calculated with higher scores reflecting worse olfactory-specific quality of life. For the sQOD-NS questionnaire composed of 7 items, the total scores range from 0 to 21.
Changes in dyspnea scale over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via modified Medical Research Council (mMRC) dyspnoea scale. | Baseline, 4 weeks, 8 weeks, 12 weeks
  The mMRC scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 m or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing.
Change in scale of Asthenia over time-point (baseline, 4 weeks, 8 weeks, 12 weeks) via asthenia scale. | Baseline, 4 weeks, 8 weeks, 12 weeks
  Analog scale from 0 to 100 mm
Change in Fatigue scale over time-point (baseline, 4 weeks, 8 weeks, 12 weeks) via Krupp Clader CFQ-11 Fatigue Intensity Scale. | Baseline, 4 weeks, 8 weeks, 12 weeks
  The Chalder Fatigue Questionnaire (CFQ) also referred to as the Chalder Fatigue Scale, is an 11-item questionnaire measuring the severity of physical and mental fatigue on two separate subscales. Seven items represent physical fatigue (items 1-7) and 4 represent mental fatigue (items 8-11). Each item is scored 0-3; less than usual (0), no more than usual (1), more than usual (2) and much more than usual (3). The ratings of items are added together to calculate the total score (range=0-33). High scores represent high levels of fatigue.
Change in Emotions scale over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via Brackets RULER scale. | Baseline, 4 weeks, 8 weeks, 12 weeks
  Brackets' RULER syllabus consists of five key skills, which anyone can learn. The acronym "RULER" stands for Recognize, Understand, Label, Express, and Regulate. The first three skills allow us to practice identifying our emotions. The last two allow us to develop the necessary skills to deal with them. The RULER curriculum is about gathering information by recognizing and understanding emotions. Apply emotional intelligence to various situations.

SECONDARY OUTCOMES:
Change of Von Willebrand Factor over time-points (baseline, 4 weeks, 12 weeks, 12 weeks) via blood sample. | Baseline, 4 weeks, 8 weeks, 12 weeks
  Von Willebrand factor will be measured by an automated, highly sensitive and specific immuno-turbidimetric assay (Liatest antigenic Stago, France. VWF in %. VWF an "acute phase protein" which increases in infections (bacterial, less viral and fungi), inflammation, post-OP, malignant processes, and represent the best biomarkers as endothelial pertubation.
Change of D Dimer over time-points (baseline, 4 weeks, 12 weeks, 12 weeks) via blood sample. | Baseline, 4 weeks, 8 weeks, 12 weeks
  D Dimer (<500 ng/ml FEU) is altered in prothrombotic or thrombotic processes.plasma levels of D-Dimer will be measured by sandwich ELISA in citrated plasma (VIDAS D-Dimer, BioMerieux SA ).
Change of HS-CRP over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via blood sample. | Baseline, 4 weeks, 8 weeks, 12 weeks
  CRP (< 0,5 mg/dl) is an "acute phase protein" which increases in infections (bacterial, less viral and fungi), inflammation, post-OP, malignant processes; ultra-sensitive CRP is additionally a risk assessment marker of aterosclerosis
Change of Ferritin over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via blood sample. | Baseline, 4 weeks, 8 weeks, 12 weeks
  Ferritin (Men: 12 to 300 ng/mL Women: 12 to 150 ng/mL.) is an "acute phase protein" which increases in infections (bacterial, less viral and fungi), inflammation, post-OP, malignant processes.

OTHER OUTCOMES:
Change of the emotional state over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via Plutchik's Wheel of Emotions. | Baseline, 4 weeks, 8 weeks, 12 weeks
  Utilizing it as a two-dimensional circle lets the individual dive into the emotion wheel. This then helps them discover what primary emotions they are feeling, as well as how emotions combine to create secondary emotions like awe, remorse, aggression, optimism, etc. It suggested that people experience eight core emotions, which it arranged in opposite pairs on the wheel: sadness and joy; anger and fear; expectation and surprise; acceptance and disgust. These basic emotions can intensify, become milder, or even combine to produce any emotional state. Looking at the wheel we can notice three main characteristics: Colors: The eight emotions are arranged by colors that establish a set of similar emotions. Layers: Moving to the center of the circle intensifies the emotion, so the colors intensify as well. Relations: The polar opposite emotions are across from each other.
Change of the emotional state over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via Scale Revised by Event Impacts. | Baseline, 4 weeks, 8 weeks, 12 weeks
  The Impact of Event Scale-Revised is a 22-item scale which is rated on a 0 (not at all) to 4 (extremely) scale with respect to how distressing each item has been during the past week. The Impact of Events Scale (IES) is one of the most widely used measures of event-specific distress. The IES assesses the frequency with which respondents experience intrusive thoughts and avoidant behaviors over the past week.
Change of the emotional state over time-points (baseline, 4 weeks, 8 weeks, 12 weeks) via Mood Person Centered Approach. | Baseline, 4 weeks, 8 weeks, 12 weeks
  Person-centered therapy, also called client-centered therapy, is a form of psychotherapy that places emphasis on the client over the therapist. It empowers the client to take control of their mental health without judgment, and helps improve the client's self-awareness

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Rubilar, PhD, Principal Investigator — Universidad Nacional de la Patagonia San Juan Bosco
Locations (1):
- Hospital Donación Francisco Santojanni, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available six month after publication for six month
Access Criteria: An email to the Principal Investigator

REFERENCES:
- [Background] Gorna R, MacDermott N, Rayner C, O'Hara M, Evans S, Agyen L, Nutland W, Rogers N, Hastie C. Long COVID guidelines need to reflect lived experience. Lancet. 2021 Feb 6;397(10273):455-457. doi: 10.1016/S0140-6736(20)32705-7. Epub 2020 Dec 23. No abstract available. PMID 33357467
- [Background] Marshall M. The four most urgent questions about long COVID. Nature. 2021 Jun;594(7862):168-170. doi: 10.1038/d41586-021-01511-z. No abstract available. PMID 34108700
- [Background] COVID-19 rapid guideline: managing the long-term effects of COVID-19. London: National Institute for Health and Care Excellence (NICE); 2024 Jan 25. Available from http://www.ncbi.nlm.nih.gov/books/NBK567261/ PMID 33555768
- [Background] S.E. de M.G. y de F. (SEMG), Guía clínica para la atención al paciente long COVID/COVID persistente, (2021) 1-12
- [Background] Raveendran AV, Jayadevan R, Sashidharan S. Long COVID: An overview. Diabetes Metab Syndr. 2021 May-Jun;15(3):869-875. doi: 10.1016/j.dsx.2021.04.007. Epub 2021 Apr 20. PMID 33892403
- [Background] Barker-Davies RM, O'Sullivan O, Senaratne KPP, Baker P, Cranley M, Dharm-Datta S, Ellis H, Goodall D, Gough M, Lewis S, Norman J, Papadopoulou T, Roscoe D, Sherwood D, Turner P, Walker T, Mistlin A, Phillip R, Nicol AM, Bennett AN, Bahadur S. The Stanford Hall consensus statement for post-COVID-19 rehabilitation. Br J Sports Med. 2020 Aug;54(16):949-959. doi: 10.1136/bjsports-2020-102596. Epub 2020 May 31. PMID 32475821
- [Background] D. Barron, Bringing the Clinical Trial to the Patient, Eye Pharma. (2017)
- [Background] Rubilar T, Barbieri ES, Gazquez A, Avaro M. Sea Urchin Pigments: Echinochrome A and Its Potential Implication in the Cytokine Storm Syndrome. Mar Drugs. 2021 May 11;19(5):267. doi: 10.3390/md19050267. PMID 34064550
- [Background] Artyukov AA, Zelepuga EA, Bogdanovich LN, Lupach NM, Novikov VL, Rutckova TA, Kozlovskaya EP. Marine Polyhydroxynaphthoquinone, Echinochrome A: Prevention of Atherosclerotic Inflammation and Probable Molecular Targets. J Clin Med. 2020 May 15;9(5):1494. doi: 10.3390/jcm9051494. PMID 32429179
- [Background] Nabavi N. Long covid: How to define it and how to manage it. BMJ. 2020 Sep 7;370:m3489. doi: 10.1136/bmj.m3489. No abstract available. PMID 32895219
- [Background] Mahase E. Long covid could be four different syndromes, review suggests. BMJ. 2020 Oct 14;371:m3981. doi: 10.1136/bmj.m3981. No abstract available. PMID 33055076
- [Background] Altmann DM, Boyton RJ. Decoding the unknowns in long covid. BMJ. 2021 Feb 4;372:n132. doi: 10.1136/bmj.n132. No abstract available. PMID 33541867
- [Background] Del Rio C, Collins LF, Malani P. Long-term Health Consequences of COVID-19. JAMA. 2020 Nov 3;324(17):1723-1724. doi: 10.1001/jama.2020.19719. No abstract available. PMID 33031513
- [Background] P. Brito-Zerón, L. Conangla Ferrín, B. Kostov, A. Moragas Moreno, M. Ramos-Casals, E. Sequeira Aymar, A. Sisó Almirall, Manfestaciones persistentes de la COVID-19 . Guía de práctica clínica, 2020.
- [Background] A.A. Artyukov, A.M. Popov, A. V. Tsybulsky, O.N. Krivoshapko, N. V. Polyakova, Pharmacological activity of echinochrome a alone and in the biologically active additive Timarin, Biochem. Suppl. Ser. B Biomed. Chem. (2013). https://doi.org/10.1134/S1990750813030025.
- [Background] N. Vinod, Living with 'Long COVID-19': The long-term complications and sequelae, Int. J. Clin. Virol. 5 (2021) 011-021. https://doi.org/10.29328/journal.ijcv.1001030.
- [Background] A.N. Shikov, O.N. Pozharitskaya, A.S. Krishtopina, V.G. Makarov, Naphthoquinone pigments from sea urchins: chemistry and pharmacology, Phytochem. Rev. (2018). https://doi.org/10.1007/s11101-018-9547-3
- [Background] C.S. Yoon, H.K. Kim, N.P. Mishchenko, E.A. Vasileva, S.A. Fedoreyev, O.P. Shestak, N.N. Balaneva, V.L. Novikov, V.A. Stonik, J. Han, The protective effects of echinochrome A structural analogs against oxidative stress and doxorubicin in AC16 cardiomyocytes, Mol. Cell. Toxicol. (2019). https://doi.org/10.1007/s13273-019-0044-6
- [Background] I.A. González, Experiencia del paciente afectado por COVID-19 persistente acerca de la utilidad y características de las escalas de valoración clínica de los síntomas derivados de su enfermedad, Med. Gen. y Fam. 9 (2020) 121-125. https://doi.org/0.24038/mgyf.2021.018.
- [Background] C.R. Rogers, Client-centered/person-centered approach to therapy, Vopr. Psikhol. (2001).
- [Background] M. Méndez, Carl Rogers y Martin Buber: las actitudes del terapeuta Centrado en la Persona y la relación " Yo-Tú " en psicoterapia, Apunt. Psicol. 32 (2014) 171-180.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT05531019/Prot_ICF_000.pdf